CLINICAL TRIAL: NCT02901756
Title: A Combination of Coenzyme Q10, Feverfew and Magnesium for Migraine Prophylaxis : a Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: PiL-Obs-AntMIG-014
Record Dates: First submitted 2016-08-24; First posted 2016-09-15 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Antemig — Participants were instructed to take one tablet every morning for three months.

SUMMARY:
Adult patients suffering from migraine according to the criteria of the International Headache Society were enrolled by general practitioners (≥2 migraine attacks during previous month; exclusion of chronic migraine and medication overuse) and after a one-month baseline phase, supplemented with one tablet of 100 mg feverfew, 100 mg coenzyme Q10 and 112.5 mg magnesium per day for 3 months.

DETAILED DESCRIPTION:
Three visits were planned: V1, V2 on Day 30 (± 10) and V3 on Day 120 (± 10). On V1, after checking the inclusion criteria and receiving informed consent, GPs collected demographic data, medical and migraine history and information on migraine attacks, associated symptoms and rescue medications via an electronic case report form. V1 was followed by a one-month observation period (baseline phase) during which migraine treatment of patients was not modified. From V1 till the end of the study, all patients kept an electronic diary in which they reported migraine characteristics (number of days with migraine headache, intensity, associated symptoms and concomitant medications). On the second visit (V2; Day 30 ± 10), eligibility of patients was verified: patients with less than 2 or more than 15 migraine attacks during baseline phase and patients unwilling to be supplemented with the combination were excluded from the study. Eligible patients were advised to start supplementation. On V3 (Day 120 ± 10), information provided in patient's diary and compliance with supplementation were checked.

The day before V2 and V3, patients had to complete the French migraine-related quality of life questionnaire (Qualité de Vie et Migraine [QVM]) and the Hospital Anxiety and Depression Scale (HADS).

The study was conducted in accordance with articles L.1121-1 and R1121-2 of the French public health code defining non interventional studies; all the acts were practised and products used in a usual way without any additional or unusual procedure of diagnosis or surveillance.

ELIGIBILITY:
Inclusion Criteria:

* to suffer from migraine with or without aura diagnosed according to the criteria of the International Classification of Headaches Disorders III (ICHD III 1.1 and 1.2)
* to suffer from migraine for more than one year
* to be less than 50 years old at migraine onset
* to have had at least two migraine attacks during the month before recruitment

Exclusion Criteria:

* migraine with aura with motor symptoms (hemiplegic migraine)
* more than 15 migraine attacks per month
* abuse of painkillers defined as the use of paracetamol, aspirin and non-steroid anti-inflammatory drugs for more than 15 days per month over the last three months or the use of triptans, opioids and ergot-type medications for more than 10 days per month during the last three months
* prophylactic treatment taken for less than 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients were recruited by general practitioners (GPs). Patients had to suffer from migraine with or without aura diagnosed according to the criteria of the International Classification of Headaches Disorders III (ICHD III 1.1 and 1.2)
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
the number of days with migraine headache at the 3rd Month | 3rd month of supplementation

SECONDARY OUTCOMES:
Number of days with migraine headache per month | during the 1st month
Number of days with migraine headache per month | during the 3rd month
Intensity of migraine headache evaluated with a 5 points Likert Scale | during the 1st month
Intensity of migraine headache evaluated with a 5 points Likert Scale | during the 3rd month
Associated symptoms evaluated with Scorecard of potential symptoms | during the 1st month of observation, 1st, 2nd and 3rd month
Associated symptoms evaluated with Scorecard of potential symptoms | during the 1st month
Anxiety and depression evaluated with DNS (Dopa Nora Sero) questionnaire | during the 3rd month
Quality of life evaluated with the QVM (Quality of Life for Migraine) questionnaire | baseline
Quality of life evaluated with the QVM (Quality of Life for Migraine) questionnaire | end of the 3rd month
Compliance followed with patient logbook | 3 months
Safety followed with side effects register | 3 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guilbot A, Bangratz M, Ait Abdellah S, Lucas C. A combination of coenzyme Q10, feverfew and magnesium for migraine prophylaxis: a prospective observational study. BMC Complement Altern Med. 2017 Aug 30;17(1):433. doi: 10.1186/s12906-017-1933-7. PMID 28854909